CLINICAL TRIAL: NCT01300494
Title: Bifurcation Optimal Viewing Angle Selection Study
Brief Title: BOVAS: Bifurcation Optimal Viewing Angle Selection Study
Acronym: BOVAS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Gasthuisberg (Other)
Collaborators: KU Leuven (Other)
Responsible Party: dr. Tom Adriaenssens, University Hospitals Leuven
Other Study IDs: BOVAS 2 08.02.2011
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Coronary Bifurcation Lesion
Keywords: bifurcation lesion; optimal viewing angle; automated software

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
An optimal angiographic viewing angle is critical for correct diagnosis and intervention in coronary bifurcation lesion percutaneous coronary interventions (PCI). The current study aims at validating a dedicated software tool (MEDIS, Leiden, The Netherlands) that will improve the selection of the best viewing angle.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years of age
* Informed consent available

Exclusion Criteria:

* Hemodynamic unstability (cardiogenic shock, life-threatening arrhythmias, inotropic support)
* Impaired renal function (serum creatinine > 2.0 mg/dl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In patients undergoing coronary angiography, those with an angiographically significant bifurcation lesion will be identified. A total of 50 patients will be selected. After diagnostic angiography, optimal viewing angles for the bifurcation lesion will be calculated using the dedicated Medis (Leiden, the Netherlands) software.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)